CLINICAL TRIAL: NCT04280731
Title: Impact of Quinoa Milk Fermented With Lactic Acid Bacteria From Foods on Human Oral and Intestinal Flora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Swedish International Development Cooperation Agency (SIDA) (Other Government)
Responsible Party: Principal Investigator, Åsa Håkansson, Principal Investigator, Lund University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FermCH
Record Dates: First submitted 2019-12-04; First posted 2020-02-21 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fermented drink (Experimental)
  Interventions: Dietary Supplement: fermented quinoa

INTERVENTIONS:
Dietary Supplement: fermented quinoa — Quinoa drink fermented with lactic acid bacteria isolated from food

SUMMARY:
The demand for alternatives to dairy products has increased in recent years and a lot of proposals for vegetable milk and yogurt products have taken place in the market. Quinoa is a plant from South America that has growth in popularity in recent years as many sought out nutritious and healthier eating, the herb is known for its high nutritional value. It is complete protein source containing all the essential amino acids. If this herb were fermented with probiotic bacteria, there is a potential for a product that is lactose free, gluten free and cholesterol free.

The probiotic potential of quinoa milk, fermented with food associated lactic acid bacteria will be investigated. This includes a study that examines how daily consumption of this vegetable drink changes the composition of the oral and intestinal flora. Therefore, healthy people are now seeking to participate in the study, which will be for just over 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years and healthy volunteers

Exclusion Criteria:

* Participants that have any kind of diseases, such as colon inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Survivability of the lactic acid bacteria | 2 weeks
  If the bacteria can be isolated in a adequate amount by cultivation on MRS broth and rogosa agar

SECONDARY OUTCOMES:
Changes in the human microbiota | 2 weeks
  Changes in the saliva and stool samples by analyzes with Terminal Restriction Fragment Length polymorphism
Changes in the human microbiota | 2 weeks
  Changes in the saliva and stool samples by quantitative polymorphic chain reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Kemicentrum, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No